CLINICAL TRIAL: NCT06787378
Title: The Sweet Dreams Study - Accuracy of Sleep Trackers in Children
Status: Recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 275668
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-01

CONDITIONS: Sleep
Keywords: sleep; accelerometer; polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children: Children ages 2 to <18 years of age will be enrolled

SUMMARY:
The study aims to evaluate the accuracy of sleep trackers in children aged 2 to less than 18 years. Children undergoing polysomnography, the gold standard for assessing sleep quality and duration, at Arkansas Children's Hospital may be eligible to participate. Participants will be asked to wear sleep trackers on the day of their sleep test. The data collected from the sleep trackers will be compared with the polysomnography results to determine the devices' accuracy.

DETAILED DESCRIPTION:
Participants will meet the research team at Arkansas Children's Hospital (ACH) two to three hours before their scheduled sleep test and are required to bring a stool sample from the child to the visit.

During the visit, the research team will gather information about the child's home environment and medical history, including parent marital status, parental education level, household income, and other factors. Questionnaires will also cover topics such as the child's growth and development, diet, physical activity, use of substances like tobacco and alcohol, and mood. Any questions that cause discomfort may be skipped by the child or their parent.

A brief physical exam will be conducted to measure the child's weight, height, blood pressure, and heart rate. Sleep trackers will then be programmed and placed, with two worn on the wrist and two around the waist. Instructions on how to remove and reattach the trackers will be provided to ensure proper use.

After completing the sleep test at ACH, the sleep trackers must be left in the sleep clinic. All four trackers must be returned, and parents will be asked to report if the trackers were removed at any point during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to <18 years
* All BMIs
* Scheduled at PSDC for evaluation of obstructive sleep apnea, snoring, or noisy breathing during sleep.

Exclusion Criteria:

* Known diagnosis of sleep disorder
* Neurological disorders (e.g., epilepsy, cerebral palsy, etc.)
* Autism spectrum disorder
* Attention deficit hyperactivity disorder
* Oppositional defiant disorder
* Chronic kidney disease
* Hormonal disease
* Autoimmune diseases
* Bleeding disorders
* Chronic infections (e.g., HIV, hepatitis B)
* Mental health disorders (e.g., depression, anxiety)
* Liver disease (e.g. hepatitis)
* Referral for evaluation of disorders other than obstructive sleep apnea, snoring, or noisy breathing during sleep.
* Pre-existing medical conditions or medications as determined by the investigators to affect the outcomes of interest.
* Refusal to authorize study investigators to access data from the polysomnography test conducted at the Arkansas Children's Hospital PSDC.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 2 to < 18years
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Total sleep time | Up to 10 days after consent
  sleep minutes between lights off and lights on
Wake after sleep onset | Up to 10 days after consent
  wake minutes between PSG-scored sleep onset and lights on
Sleep efficiency | Up to 10 days after consent
  Total sleep time divided by sleep period or number of total min from lights off to lights on

CONTACTS AND LOCATIONS:
Overall Officials: Eva C Diaz, MD, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Arkansas Children's Nutrition Center, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: Yes
study protocol, and consent, analytic code
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: upon publication of primary outcomes of interest
Access Criteria: Researchers affiliated with recognized academic institutions who propose scientifically valid research questions.
  Researchers will submit a data access request, including a study proposal, objectives, and intended use of the data.
  Approval will be determined by a data-sharing committee or equivalent oversight body.

REFERENCES:
- [Background] Lu MJ, Zhong WH, Liu YX, Miao HZ, Li YC, Ji MH. Sample Size for Assessing Agreement between Two Methods of Measurement by Bland-Altman Method. Int J Biostat. 2016 Nov 1;12(2):/j/ijb.2016.12.issue-2/ijb-2015-0039/ijb-2015-0039.xml. doi: 10.1515/ijb-2015-0039. PMID 27838682
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Smith C, Galland B, Taylor R, Meredith-Jones K. ActiGraph GT3X+ and Actical Wrist and Hip Worn Accelerometers for Sleep and Wake Indices in Young Children Using an Automated Algorithm: Validation With Polysomnography. Front Psychiatry. 2020 Jan 14;10:958. doi: 10.3389/fpsyt.2019.00958. eCollection 2019. PMID 31992999
- [Background] Quante M, Kaplan ER, Cailler M, Rueschman M, Wang R, Weng J, Taveras EM, Redline S. Actigraphy-based sleep estimation in adolescents and adults: a comparison with polysomnography using two scoring algorithms. Nat Sci Sleep. 2018 Jan 18;10:13-20. doi: 10.2147/NSS.S151085. eCollection 2018. PMID 29403321